CLINICAL TRIAL: NCT04743362
Title: Noninvasive Assessment of Muco-cutaneous Lesions In Vivo
Brief Title: A Study of Noninvasive Methods to Evaluate Skin and Mucosal Conditions
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-019
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Skin Lesion; Mucosal Lesion
Keywords: muco-cutaneous lesion; skin lesion; mucosal lesion; Memorial Sloan Kettering Cancer Center; 21-019
MeSH Terms: interventions — Microscopy, Confocal; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with muco-cutaneous lesions: Participants will have muco-cutaneous lesions for non-invasive evaluation (including normal skin or mucosa and benign lesions) and will be identified by their physicians or fellows during routine clinical care.
  Interventions: Diagnostic Test: Dermoscopic imaging; Diagnostic Test: 3-dimensional total body photography; Diagnostic Test: Confocal microscopy; Diagnostic Test: Optical Coherence Tomography imaging; Diagnostic Test: Ultrasound; Diagnostic Test: Hyperspectral imaging; Diagnostic Test: Electrical impedance spectroscopy; Diagnostic Test: Patient self-imaging

INTERVENTIONS:
Diagnostic Test: Dermoscopic imaging — The skin lesion will be imaged before application of alcohol (spray/wipe) and after application of alcohol (spray/wipe). The dermatoscope/camera with dermoscopy imaging capabilities, including but not limited to VEOS® SLR (Canfield Scientific, Inc.), will be placed on/near the area(s) of interest. Images will be captured in polarized and/or nonpolarized modes and contact and/or non-contact modes.
Diagnostic Test: 3-dimensional total body photography — Participants will stand in the center of an imaging station consisting of 92 high-resolution cameras. Image capture by all cameras will occur simultaneously, (approx. 3 milliseconds). Within a few minutes, specialized software will process and assemble the images into a 3D avatar - a digital model of the patient's skin - showing all his or her lesions.
  Other Names: 3D TBP
Diagnostic Test: Confocal microscopy — CM imaging (Vivascope®, Caliber Imaging and Diagnostics, Rochester, NY) will be performed using an arm-mounted CM device (Vivascope1500, Caliber I.D., Inc.) or using a handheld CM device (Vivascope3000, Caliber I.D., Inc.).
  Other Names: CM
Diagnostic Test: Optical Coherence Tomography imaging — OCT subsurface imaging shows structural-level morphology (epidermal and dermal layers) in skin down to the deeper reticular dermis.
  Other Names: OCT imaging
Diagnostic Test: Ultrasound — US imaging allows assessment of depth, Doppler vascular imaging, and elastography features of skin lesions.
  Other Names: US
Diagnostic Test: Hyperspectral imaging — Hyperspectral imaging shows biochemical information regarding the distribution of skin melanin and hemoglobin50. SkinSpect™ is a form of a hyperspectral dermatoscope.
Diagnostic Test: Electrical impedance spectroscopy — Electrical impedance spectroscopy (EIS) measures skin's resistance to the flow of alternating electric currents to differentiate benign and malignant lesions.
  Other Names: EIS
Diagnostic Test: Patient self-imaging — Clinical and dermoscopy self-imaging by patients can be accomplished using mobile phone technology. In the case of dermoscopy, this requires a small dermatoscope attachment for the phone.

SUMMARY:
The purpose of this study is to find out whether using noninvasive methods to study the appearance of lesions can improve diagnostic accuracy before a biopsy is required and help guide treatment planning. The database created to store these images is called an Image Repository, and it will be used to support clinical practice, teaching and training, and future research.The High-resolution OCT (Apollo Medical Optics) device ApolloVue® S100 Image System (medical device Class II) can provide both cross-sectional and en-face images with cellular information.

ELIGIBILITY:
Inclusion Criteria:

* All ages
* Patients with a muco-cutaneous lesion(s) amenable to imaging by non-invasive tools
* Healthy volunteer subjects
* Ability to give informed consent or in the case of pediatric patients, assent and consent from the parent/guardian

Exclusion Criteria:

* Allergy or intolerance to ultrasound gel or mineral oil used for imaging
* Patients who are not able to comply with imaging procedure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For this study, we anticipate to recruit ~5000 participants over a period of 7 years. Of this, ~4000 will be patients with a muco-cutaneous lesion and ~1000 will be volunteers.
  Patients in the Dermatology, Clinical Immunology Services, Pediatrics, Bone Marrow Transplant, Dental, and Radiation Oncology departments who have a muco-cutaneous lesion/process amenable to imaging with one or more of the available noninvasive devices will be offered the opportunity to participate in the study. In addition to patients and volunteers, MSK clinicians will be recruited to the study via clinician verbal informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 5010 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2031-08-02 (Estimated); Study Completion 2031-08-02 (Estimated)

PRIMARY OUTCOMES:
Collect images of untreated and treated neoplastic and non-neoplastic muco-cutaneous conditions | 7 years
  The primary outcome of this study is to collect images from varied images devices with the dermatology service and to create an effective mechanism for the storage and dissemination of the resultant images for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Manu Jain, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org